CLINICAL TRIAL: NCT04433533
Title: A Randomized, Single-center, Open, Parallel, Phase 4 Study to Compare the Efficacy and Safety of Rosuvastatin/Ezetimibe Combination Therapy Versus Rosuvastatin Monotherapy in Korean Patients With Left Ventricular Diastolic Dysfunction and Hyperlipidemia
Brief Title: Compare the Efficacy and Safety of Rosuvastatin/Ezetimibe Combination Therapy Versus Rosuvastatin Monotherapy in Korean Patients With Left Ventricular Diastolic Dysfunction and Hyperlipidemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1125
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Left Ventricular Diastolic Dysfunction; Hyperlipidemias
MeSH Terms: conditions — Ventricular Dysfunction, Left; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin 20mg (Group 1) (Active Comparator)
  Interventions: Drug: Rosuvastatin 20
- Rosuvamibe 10/10mg (Group 2) (Experimental)
  Interventions: Drug: Rosuvamibe 10/10

INTERVENTIONS:
Drug: Rosuvastatin 20 — Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of Rosuvastatin 20mg Monotherapy.
  Arms: Rosuvastatin 20mg (Group 1)
Drug: Rosuvamibe 10/10 — Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly enrolled in a 1: 1 dose of rosuvastatin10mg/ezetimibe 10mg combination Therapy
  Arms: Rosuvamibe 10/10mg (Group 2)

SUMMARY:
preserved left ventricular ejection fraction (LVEF ≥ 50%) and are accompanied by dyslipidemia (LDL ≥ 100 mg / dl) will be enrolled.

Only patients who do not meet the exclusion criteria should be enrolled in the study.

Once the patient is selected, the patient is informed of the study and receives the consent form.

Patients who are eligible for all of the criteria and who do not qualify as exclusion criteria should be enrolled in the study and randomly assigned in a 1: 1 dose of rosuvastatin/ezetimibe 10/10mg once daily or rosuvastatin 20 mg once daily. Patients who previously used statins have a wash-out period of 4 weeks or more.

Patients will visit outpatient clinic at 12 weeks and 24 weeks after initiation of treatment. Physical examination, blood test, and 6 minute working test will be performed. For fasting blood tests, patients visit on an empty stomach. Drug adverse events and changes in vital signs or body weight will be checked.

After 48 weeks of treatment, the patients will visit outpatient clinic for efficacy evaluation; physical examination, blood test, transthoracic echocardiography, cardiopulmonary exercise test, central blood pressure, and pulse wave velocity. Drug adverse events and medication compliance will be checked.

The primary endpoint is change of low-density lipoprotein cholesterol and secondary endpoint is improvement of diastolic dysfunction, VAC index, peak VO2, distance of 6 minute working test, and clinical outcomes including death, readmission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have left ventricular diastolic dysfunction (relaxation abnormality, pseudonormalization, restrictive pattern) with preserved left ventricular systolic function (left ventricular ejection fraction ≥ 50%)
2. Adult participants (≥ 20 years old) who have dyslipidemia and need treatment
3. Patients who understand the information about the trial and voluntarily agree to participate in the trial

Exclusion Criteria:

1. Baseline fasting low-density lipoprotein cholesterol ≤ 70 mg/dL
2. Baseline fasting triglyceride ≥ 400 mg/dL
3. Baseline fasting total cholesterol ≥ 300 mg/dL
4. Participants who have structural heart disease
5. Participants who have prior acute coronary syndrome or cerebrovascular attack within 3 months.
6. Renal dysfunction (estimated glomerular filtration rate < 30mL/min/1.73m2)
7. Creatinine phosphokinase elevations greater than three times the upper limit of normal
8. Aspartate or alanine aminotransferase elevations greater than three times the upper limit of normal
9. Previous history of rhabdomyolysis
10. Females who are pregnant or breastfeeding or have a plan for pregnancy
11. Life expectancy less than a year.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum level of low-density lipoprotein cholesterol | 24 weeks
  Compare the evaluation low-density lipoprotein cholesterol changes in Rosuvastatin/Ezetimibe Combination Therapy versus Rosuvastatin Monotherapy
Change in serum level of low-density lipoprotein cholesterol | 48 weeks
  Compare the evaluation low-density lipoprotein cholesterol changes in Rosuvastatin/Ezetimibe Combination Therapy versus Rosuvastatin Monotherapy

SECONDARY OUTCOMES:
Improvement of diastolic dysfunction | 48 weeks
Improvement of ventriculoarterial coupling index | 48 weeks
Improvement of peak VO2 | 48 weeks
Improvement of 6 minute walking test combination therapy and monotherapy | 48 weeks
Clinical outcomes including death rate | 48 weeks
Clinical outcomes including readmission rate | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No